CLINICAL TRIAL: NCT07062419
Title: The Effects of Sonic Activation of Irrigant on Post Operative Pain After Root Canal Treatment on Permanent Dentition: A Randomized Clinical Study
Brief Title: Effect of Sonic Activation of Irrigant on Post Operative Pain After Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Responsible Party: Principal Investigator, Samia Rasool, Principal Investigator, CMH Lahore Medical College and Institute of Dentistry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107/Civ/Trg/Op/15/24
Record Dates: First submitted 2025-06-20; First posted 2025-07-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-06

CONDITIONS: Post Operative Pain; Root Canal Therapy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- one group will receive irrigation during root canal treatment will be activated by an Endoactivator (Experimental): activation of an irrigant by using certain ultrasonic frequency to enhance antimicrobial action of irrigant
  Interventions: Device: endoactivator
- One group will receive irrigation during root canal treatment in which activation will not occur (No Intervention): This group consists of patients who will receive irrigation during root canal treatment using the conventional syringe irrigation technique without the use of the EndoActivator system.

INTERVENTIONS:
Device: endoactivator — activation of irrigant during root canal treatment
  Arms: one group will receive irrigation during root canal treatment will be activated by an Endoactivator

SUMMARY:
Fifty-eight patients aged 18-60 years, diagnosed with symptomatic or asymptomatic apical periodontitis will be randomly allocated into two groups: Group A (EndoActivator) and Group B (conventional syringe irrigation). preoperative pain will be evaluated in all patients requiring root canal treatment using visual analogue scale before initiating the procedure.

Postoperative pain will be measured using the Visual Analog Scale (VAS) at 24, 36, 48 hours and one week.

DETAILED DESCRIPTION:
This randomized clinical study will evaluate the effect of two different irrigation techniques on postoperative pain following root canal treatment in patients with apical periodontitis. A total of 58 patients will be randomly assigned to one of two groups: one group will receive irrigation using the EndoActivator system, while the other group undergo conventional syringe irrigation. The objective is to determine whether the irrigation technique influences the level of postoperative discomfort experienced by patients. Pain levels will be assessed at specific time intervals to track the pattern of recovery and provide insight into the clinical effectiveness of each method in terms of patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* irreversible pulpitis
* symptomatic apical periodontitis
* asymptomatic apical periodontitis
* compliant patients
* sufficient ferrule for post operative restoration

Exclusion Criteria:

* periapical abcess
* severe periodontal disease with guarded periodontal prognosis
* teeth with guarded post operative restoration prognosis
* non compliant patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
post operative pain using endoactivator | before procedure, after 24 hours, 36 hours , 48 hours, 1 week
  post operative pain will be marked on visual analogue scale (VAS). the lower the score the less pain will be and vice versa.
  maximum score 10 minimum score 0 0 to 10 depicting no pain to worst pain
post operative pain | before procedure, after 24 hours , 36 hours , 48 hours , 1 week
  pain will be evaluatedon visual analogue scale (VAS). the lower the score the less pain will be and vice versa.
  maximum score 10 minimum score 0 0 to 10 depicting no pain to worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Imran Khan, BDS FCPS, Study Director — 28 military dental centre
Locations (1):
- 28 Military Dental Centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No